CLINICAL TRIAL: NCT01556191
Title: Phase II Randomised Clinical Trial Evaluating an EGFR Tyrosine Kinase Inhibitor (EGFR-TKI) Versus an EGFR-TKI Combined With an Anti-oestrogen Treatment (Fulvestrant) in Women With Advanced Stage Non-squamous Lung Cancer
Brief Title: Lung Cancer in Women Treated With Anti-oestrogens anD Inhibitors of EGFR
Acronym: LADIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1003
Record Dates: First submitted 2012-03-08; First posted 2012-03-16 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Stage IV Lung Cancer
Keywords: lung cancer; women
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib; Fulvestrant; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gefinitib + Fulvestrant (patient with EGFR mutations) (Experimental)
  Interventions: Drug: Gefitinib; Drug: Fulvestrant
- Erlotinib (wild type patients) (Active Comparator)
  Interventions: Drug: Erlotinib
- Erlotinib + Fulvestrant (wild type patients) (Experimental)
  Interventions: Drug: Fulvestrant; Drug: Erlotinib
- Gefinib (patient with EGFR mutations) (Active Comparator)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250 mg per day (oral)
  Arms: Gefinib (patient with EGFR mutations); Gefinitib + Fulvestrant (patient with EGFR mutations)
Drug: Fulvestrant — 500 mg (2 x 250 mg), IV by month with an additional 500 mg dose two weeks after the initial dose
  Arms: Erlotinib + Fulvestrant (wild type patients); Gefinitib + Fulvestrant (patient with EGFR mutations)
Drug: Erlotinib — 150 mg per day (oral)
  Arms: Erlotinib (wild type patients); Erlotinib + Fulvestrant (wild type patients)

SUMMARY:
Lung Cancer is to become the first cause of death related to cancer in France as it's already the case in United States. At Present, Lung Cancer in women and in men is treated similarly. Nevertheless, numerous studies shows that lung cancer in women has specificities : at the time of the diagnosis female patients are younger, there are less clinical signs, clinical stages are earlier, histology is often adenocarcinoma. The link with tabagism is weaker . Sensitivity to tabagism is higher (more cancer in women with the same tabagism). Response rate to chemotherapy is better. Prognosis is better

Numerous hypotheses have been put forward to account for the specific characteristics of female lung cancer described above.

* One hypothesis is that there are different genetic anomalies in women. Some studies show an increase of EGFR mutation and HER2 expression and a decrease of expression of repair enzymes (ERCC1, RRM1, BRCA) which can explain the increase sensitivity to tabagism and to chemotherapy.
* Another hypothesis is that hormones play a role in oncogenesis. Indeed, lung cancer presents hormonal risk factors : pre-menopause, less than 3 kids, short menstrual cycle, hormone replacement therapy. Estrogens would have a deleterious effect on cancer incidence and on survival of lung cancer in women. Cellular and animal models show that ER pathway is activated in lung cancer and participates in oncogenesis.
* Moreover an interaction between RE and EGFR pathway has been demonstrated on lung cancer cell lines and mouse models.

EGFR-TKI have shown benefit in women with wild type EGFR or unknown status (with erlotinib) and in women with EGFR mutations (with gefitinib). In this study, the use of these two treatment will be in accordance with their market authorisations.

The objective of this study is to test the addition of an anti-estrogen (fulvestrant) to EGFR-TKI. Fulvestrant is a pure anti-oestrogen that binds to ER, blocks it and accelerates its breakdown. It has a market authorisation in breast cancer. Furthermore the association between EGFR-TKI and anti-estrogen could have a synergetic effect due to interaction between RE and EGFR pathways .

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed predominant non-squamous, non-small cell lung cancer
* The presence of analysable tissue for the research of EGFR activating mutation. Analysis must be performed in INCa-labelled laboratories or platforms according to a validated technique
* Not suitable for radiation, inoperable stage III or stage IV
* Patients with an EGFR mutation must never have taken chemotherapy or must be in progression after only one previous line of chemotherapy (including maintenance). Patients without an EGFR mutation must have received one or two lines of chemotherapy beforehand. Maintenance chemotherapy is not considered to be a treatment line. Adjuvant chemotherapy is not considered to be a first line of treatment if it dates back to over a year
* Female
* Menopausal: older than 60 years of age or history of ovariectomy or younger than 60 years old with amenorrhoea for more than 12 months or an FSH rate that corresponds to a post-menopausal rate (according to the laboratory)

Exclusion Criteria:

* History of cancer except for skin cancer or cancer dating from over five years ago and considered to be cured
* Known or suspected Cerebral metastases or spinal cord compression unless they are asymptomatic without treatment or stable after being treated by surgery and/or radiation therapy. Corticosteroid treatments for symptoms must have discontinued for more than four weeks
* Pregnancy and breast-feeding
* Patient taking hormone replacement therapy for menopause that has not been stopped two weeks before the start of the trial treatment
* A change in bone marrow, kidney and liver functions inconsistent with treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
progression-free survival | Around nine months
  From date of randomization until the date of first progression for EGFR mutated patient
Progression free survival | Around three months
  From date of randomization until the date of first progression for EGFR wild type patients

SECONDARY OUTCOMES:
toxicity of EGFR-TKI and fulvestrant | Around three months
  The number of patients for whom at least an adverse event will have been reported, the number of events, according to the relation to the treatment, the intensity, and the cycle of appearance for EGFR WT patients
Response rate | Around three months
  For EGFR WT patients
Overall survival | Up to 18 months
  For all patients
toxicity of EGFR-TKI and fulvestrant | Around Nine months
  The number of patients for whom at least an adverse event will have been reported, the number of events, according to the relation to the treatment, the intensity, and the cycle of appearance for EGFR mutated patients
Response rate | Around nine months
  For EGFR-Mutated patients

CONTACTS AND LOCATIONS:
Overall Officials: Julien MAZIERES, MD, phD, Principal Investigator — University Hospital, Toulouse
Locations (61):
- France (61):
  - Annemasse - CH, Ambilly
  - Clinique de l'Europe, Amiens
  - Angers - CHU, Angers
  - CH de la Côte Basque, Bayonne
  - CHU Besancon - Pneumologie, Besançon
  - Béziers - CH, Béziers
  - Bobigny - Hôpital Avicenne, Bobigny
  - Hôpital Ambroise Paré - Pneumologie, Boulogne
  - HCL Hôpital Louis Pradel, Bron
  - Caen - Centre François Baclesse, Caen
  - Caen - CHU Côte de Nacre, Caen
  - Cahors - CH, Cahors
  - Chambéry - CH, Chambéry
  - Centre Hospitalier, Chauny
  - Hôpital de Cholet - Pneumologie, Cholet
  - Clamart - Hôpital Percy, Clamart
  - CHU, Clermont-Ferrand
  - CH, Colmar
  - Clinique des Cèdres, Cornebarrieu
  - Créteil - CHI, Créteil
  - CH de Dax, Dax
  - Dijon - CAC, Dijon
  - Grenoble - CHU, Grenoble
  - Chartres - CH, Le Coudray
  - Centre Hospitalier - Pneumologie, Le Mans
  - CHU (Hôpital Calmette) - Pneumologie, Lille
  - CH, Longjumeau
  - Hôpital Nord - Oncologie Multidisciplinaire & Innovations Thérapeutiques, Marseille
  - Institut Paoli Calmette, Marseille
  - Polyclinique du Val de Sambre, Maubeuge
  - Mont de Marsan - CH, Mont-de-Marsan
  - Mulhouse - CH, Mulhouse
  - CHU Nancy, Nancy
  - Nantes - Centre René Gauducheau, Nantes
  - Nevers - CH, Nevers
  - Centre Antoine Lacassagne, Nice
  - Hopital Tenon - Pneumologie, Paris
  - HIA Val-de-Grâce, Paris
  - Hôpital Bichat - Claude - Bernard, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint-Joseph, Paris
  - Paris - Curie, Paris
  - Pau - CH, Pau
  - Perpignan - Ch, Perpignan
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Centre Hospitalier, Rambouillet
  - CHU de Reims, Reims
  - Institut Jean Godinot, Reims
  - Rouen - CHU, Rouen
  - Saint Quentin - CH, Saint-Quentin
  - Strasbourg - NHC, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Centre Hospitalier Intercommunal, Toulon
  - Clinique Pasteur, Toulouse
  - Toulouse - CHU Larrey, Toulouse
  - Tourcoing - CH, Tourcoing
  - CHU Tours - Pneumologie, Tours
  - Versailles - CH, Versailles
  - CHI de la Haute-Saône - Pneumologie, Vesoul
  - CH de Villefranche - Pneumologie, Villefranche
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Mazieres J, Barlesi F, Rouquette I, Molinier O, Besse B, Monnet I, Audigier-Valette C, Toffart AC, Renault PA, Fraboulet S, Hiret S, Mennecier B, Debieuvre D, Westeel V, Masson P, Madroszyk-Flandin A, Pichon E, Cortot AB, Amour E, Morin F, Zalcman G, Moro-Sibilot D, Souquet PJ. Randomized Phase II Trial Evaluating Treatment with EGFR-TKI Associated with Antiestrogen in Women with Nonsquamous Advanced-Stage NSCLC: IFCT-1003 LADIE Trial. Clin Cancer Res. 2020 Jul 1;26(13):3172-3181. doi: 10.1158/1078-0432.CCR-19-3056. Epub 2020 Mar 6. PMID 32144133
- See also: IFCT official website — http://www.ifct.fr